CLINICAL TRIAL: NCT04454606
Title: The New Silicone N99 Half-Piece Respirator:VJR-NMU N99:New and Effective Tool to Prevent COVID-19
Brief Title: The New Silicone N99 Half-Piece Respirator
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bangkok Metropolitan Administration Medical College and Vajira Hospital (Other Government)
Responsible Party: Principal Investigator, Thananda Trakarnvanich, Associate Professor, Bangkok Metropolitan Administration Medical College and Vajira Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 053/2563
Record Dates: First submitted 2020-06-26; First posted 2020-07-01 (Actual); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: COVID; Personal Protective Equipment
Keywords: respirators; n99; COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: N99 respirators will be tested in a group of subjects with qualitative fit test.The filters will be tested for filtration test.The results will be considered as pass or fail
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fit test (Experimental): All the subjects will be tested for fit test
  Interventions: Device: Fit test; Device: Filtration Test

INTERVENTIONS:
Device: Fit test — Bitrex Fit Test The Bitrex test uses a person's ability to test a bitter solution to determine whether a respirator fits properly[11]. Each subject was given a taste-threshold screening test prior to each fit test to ensure that he or she could taste. This process was done without subject wearing a respirator. After passing the sensitivity test, the subject will process to 7 steps of fit test as following
  * Breathe normally
  * Breathe deeply
  * Head side to side
  * Head up and down
  * Bent over wrist, jogging
  * Talking
  * Breath normally Each step took 60 seconds and the Bitrex solution was refilled into the hood every 30 seconds with half dosage of the amount of the previously test. We asked the participant if he / she could taste the solution during each steps of the test . The test was considered a failure, otherwise, a pass.
Device: Filtration Test — Respirator Performance
  The real time respirator performance test method was developed using MT-05U machine (SIBATA model, Saitama, Japan), which measure particle concentrations of diameter 0.03 - 0.06 µm using and particle generator laser beam scattering particle counter that measure particles outside and inside the mask. The ratio between these two values reflected % leak as following:
  * leak=((Paticle inside the filter))/((Paticle inside the filter)) x 100 And calculate % filter performance = 100 - % leak We tested at the airflow rate of 40L/min which is 3-4 times higher than normal physiology, assuming that there should be no leakage through the filter. We tested 2 types of filter is CareStar and SafeStar that was incorporated with the silicone mask. CareStar is limited for 24 hour usage and SafeStar is for 72 hour duration.
  Study protocol

SUMMARY:
Filter facepiece respirator (FFR) is a critical equipment to prevent the transmission of respiratory tract infection disease especially the dreadful corona virus 2(SARs-CoV-2).The N95 mask is the prototype of high efficiency protective device and can effectively protect airborne pathogens of less than 0.3 μm by more than 95%. It is tightly fit and had high filtration capacity. The widespread pandemic of COVID-19 leads to greater requirement of FFR. A rising in demand would greatly exceed current productive capabilities and stockpiles and would almost certainly result in a robust shortage.

In order to solve these problems, our team had invented a new type of half-piece respirator made from silicone and assembled with hepa or elastostatic filter . A variety of methods have been used to evaluate this new device, including qualitative fit test with Bitrex® test kit and filtration test.

DETAILED DESCRIPTION:
As required by Occupational Safety and Health Administration OSHA)[7], the halfpiece respirators need to pass the fittestto identify those individuals who do not achieve the good fit necessary for adequate protection. The performance of this respirator was also determined by measuring percent leakage under constant airflow[8]. The purposes of this study was to evaluate the fitting characteristicof our newly invented silicone N99 respirator and the performance against 30 µm particles using NaCL aerosols. The study was conducted to achieve two specific research objectives

1. To investigate the fit characteristic of the novel silicone mask and whether the strap adjustment can help reduce the face-seal leakage
2. To determine the level of performance by measure the inward leakage of the generated aerosolswith the new filter and used filter for up to 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* Healthcare workers

Exclusion Criteria:

* Intolerance to exercise
* cannot taste bitter sensation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-05-15 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Fit test | Day 1
  pass or fail

OTHER OUTCOMES:
Filtration test | Day 1
  percent leakage less than1 percent

CONTACTS AND LOCATIONS:
Overall Officials: Thananda Trakarnvanich, M.D., Study Director — Bangkok Metropolitan Administration and Vajira Hospital
Locations (1):
- Bangkok Metroplitan Administration and Vajira Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gralton J, Tovey E, McLaws ML, Rawlinson WD. The role of particle size in aerosolised pathogen transmission: a review. J Infect. 2011 Jan;62(1):1-13. doi: 10.1016/j.jinf.2010.11.010. Epub 2010 Nov 19. PMID 21094184
- [Background] 5.Occupational Safety and health Administration(OSHA): 29 CFR parts 1910 and 1926 Respiratory Protection: Final Rule. Federal Register 63(5): 1278-1279. Washington, D.C: U.S. Government Printing Office, Office of the Federal Register, January 8,1998.
- [Background] Coffey C, Zhuang Z, Campbell D. Evaluation of the BitrixTM qualitative fit test method using N95 filtering-facepiece respirators. J Int Soc Respir Prot 1998: 16 : 48-55.
- [Result] Leung NHL, Chu DKW, Shiu EYC, Chan KH, McDevitt JJ, Hau BJP, Yen HL, Li Y, Ip DKM, Peiris JSM, Seto WH, Leung GM, Milton DK, Cowling BJ. Author Correction: Respiratory virus shedding in exhaled breath and efficacy of face masks. Nat Med. 2020 Jun;26(6):981. doi: 10.1038/s41591-020-0946-9. PMID 32461699